CLINICAL TRIAL: NCT06533254
Title: Use of Behavioral Artificial Intelligence to Predict and Increase Uptake of Peritoneal Dialysis [AI-Dialysis]
Brief Title: Behavioral AI to Predict and Increase Peritoneal Dialysis Uptake
Acronym: AI
Status: Recruiting | Type: Observational
Sponsor: Scaled Insights (Industry)
Collaborators: Dallas Renal Group (Unknown); The Leeds Teaching Hospitals NHS Trust (Other); Suffolk and North East Essex NHS Trust (Unknown)
Responsible Party: Principal Investigator, Stuart W. Flint, Dr Stuart W. Flint, University of Leeds
Other Study IDs: AI-Dialysis
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Artificial Intelligence; Dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients who have Chronic Kidney Disease (Phase 1): Patients who have Chronic Kidney Disease attending clinics managed by Dallas Renal Group in Texas USA, Leeds Teaching Hospitals NHS Trust UK and Suffolk and North East Essex NHS Trust UK will be contacted via their health care provider to invite them to participate.
  Interventions: Other: Predicting choice of dialysis
- Patients who have Chronic Kidney Disease (Phase 2): Patients who have Chronic Kidney Disease and are attending the units managed by Dallas Renal Group in Texas USA, Leeds Teaching Hospitals NHS Trust UK and Suffolk and North East Essex NHS Trust UK.
  Interventions: Behavioral: Behavioral nudges

INTERVENTIONS:
Other: Predicting choice of dialysis — Language data collected using survey 1, will be analyzed using Scaled Insights Behavioral AI solution to identify personality attributes and values. The resulting individual scores will be plotted on a graph and be used to identify specific personality clusters of patients.
  Participants will respond to a survey that utilizes open and closed ended questions, asking broad questions about kidney failure and associated behaviors (e.g. diet, attitudes towards treatment). The open-ended questions will gather a natural language sample of 100-300 words whilst closed questions will capture data using Likert scale and multiple-choice responses.
  The open-ended questions will gather a natural language sample of 100-300 words for analysis using Scaled Insights Behavioral AI approach. This language sample will be analyzed using Scaled Insights Behavioral AI system to identify personality attributes and values. Patients will also be asked their likelihood of selecting PD over HD.
  Groups: Patients who have Chronic Kidney Disease (Phase 1)
Behavioral: Behavioral nudges — Patients with Chronic Kidney Disease, participants will be provided with their predicted personalized nudge to increase their likelihood of either maintaining their choice of peritoneal dialysis, or switching from hemodialysis to peritoneal dialysis.
  Participants will respond to a survey that utilizes open and closed ended questions, asking broad questions about kidney failure and associated behaviors (e.g. diet, attitudes towards treatment). The open-ended questions will gather a natural language sample of 100-300 words whilst closed questions will capture data using Likert scale and multiple-choice responses.
  Groups: Patients who have Chronic Kidney Disease (Phase 2)

SUMMARY:
Scaled Insights Behavioral AI will be used to improve clinicians ability to detect and understand: The likelihood of patients with kidney failure opting for peritoneal dialysis and to select the right personalized nudge to get CKD patients to choose peritoneal dialysis

Scaled Insights' can utilize the data from this study to develop individualized nudges for healthcare professionals that can be broadly deployed within a digital platform so that clinics across the English speaking world can use it as a means of supporting patients with CKD in selecting peritoneal dialysis treatment.

Using Scaled Insights novel Behavioral Artificial Intelligence solution, the proposed project has two aims:

1. to identify personality attributes of patients with Chronic Kidney Disease and correlating their personality attributes with their subsequent choice of dialysis. Once correlated into personality based clusters, the AI Model will then be able will determine which personality cluster each net new patient will fall into and therefore predict their specific likelihood of opting for peritoneal dialysis or hemodialysis
2. once prediction is possible, customized nudges towards the selection of PD will be developed and tested to improve the likelihood that patients will opt for peritoneal dialysis

Hypotheses:

1. Scaled Insights Behavioral AI will identify the personality characteristics of patients with Chronic Kidney Disease who are likely to opt for both peritoneal dialysis and hemodialysis (Phase 1)
2. Scaled Insights Behavioral AI will identify the nudges that are most effective in encouraging or supporting patients with Chronic Kidney Disease in choosing peritoneal dialysis over hemodialysis (Phase 2)

ELIGIBILITY:
Inclusion Criteria:

* Phase 1: US and UK adult patients aged 18+ years, with Chronic Kidney Disease stage 4-5.
* Phase 2: US and UK adult patients aged 18+ years, with Chronic Kidney Disease stage 4-5.

Exclusion Criteria:

* Phase 1: Young people aged <18 years. People who do not have Chronic Kidney Disease. People who reside outside of the USA and UK.
* Phases 2: Young people aged <18 years. People who do not have Chronic Kidney Disease stage 4-5. People who reside outside of the USA and UK.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are two phases in this study.
  Phase 1: 2000 participants in total. 1000 in the USA, and 1000 in the UK; 500 patients who predict they will choose peritoneal dialysis and 500 who predict they will choose hemodialysis in each country.
  Patients who agree to participate in the study, will consent using an online survey disseminated to patients with Chronic Kidney Disease stage 4-5. Where needed, participants can be supported to complete the survey by a Research Nurse/Assistant to complete the survey.
  Phase 2: 1000 Patients with Chronic Kidney Disease in total. 500 in the USA and 500 in the UK.
  Patients who agree to participate in the study. They will be asked to access a link to an online web platform where the study will be hosted.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Choice of Dyalysis | From August 2024 to August 2025
  The Investigators will use AI to predict patients choice of dialysis. This choice will be recorded by their clinical provider as per normal routine care.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart W Flint, PhD, Principal Investigator — Scaled Insights
Locations (1):
- Dallas Renal Group, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flint SW, Brown A, Tahrani AA, Piotrkowicz A, Joseph AC. Cross-sectional analysis to explore the awareness, attitudes and actions of UK adults at high risk of severe illness from COVID-19. BMJ Open. 2020 Dec 29;10(12):e045309. doi: 10.1136/bmjopen-2020-045309. PMID 33376185
- [Background] Flint SW, Leaver M, Griffiths A, Kaykanloo M. Disparate healthcare experiences of people living with overweight or obesity in England. EClinicalMedicine. 2021 Sep 15;41:101140. doi: 10.1016/j.eclinm.2021.101140. eCollection 2021 Nov. PMID 34585130
- See also: Website for the AI company that developed the AI solution that will be used in this study. — https://www.scaledinsights.com/